CLINICAL TRIAL: NCT03896256
Title: Ketamine for Refractory Chronic Migraine: a Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Eric Schwenk, Associate Professor, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19D0.99
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Migraine Headache With Intractable Migraine
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Patients will be admitted to the hospital for a total of 5 full days from the time of admission until discharge. Ketamine infusion will be started on day 1. Adjustments to ketamine infusion will be made according to standard acute pain service protocol.
  Interventions: Drug: ketamine infusion

INTERVENTIONS:
Drug: ketamine infusion — Ketamine will be used in subanesthetic doses for patients with refractory chronic migraine to see if it improves pain after a 5-day continuous infusion.
  Other Names: Ketalar

SUMMARY:
Ketamine is a drug used for anesthesia but at low doses it is a very effective pain reliever in several chronic conditions. Preliminary studies have shown that ketamine might be effective for patients with refractory chronic migraine, which is a severe type of headache for which patients usually have tried and failed many medications and can cause severe disability to their lives. This study will evaluate ketamine prospectively when given to patients who have "failed" an initial inpatient treatment.

DETAILED DESCRIPTION:
This study is a comparison between ketamine, used in the standard fashion at Thomas Jefferson University Hospital (TJUH) for 5 days, and past data collected from inpatient treatment at Methodist Hospital. The collection of blood samples is the only experimental part of the study.

Eligible patients will be identified by a study team member at the end of inpatient treatment at Methodist Hospital. The study will be explained to patients at that time. Patients who express interest in participation will be given a consent packet to take home and bring to their office visit at Jefferson Headache Center prior to admission to TJUH for ketamine infusions. Patients will be given the time to read over the study information and have all questions answered to their satisfaction. The will provide informed consent at the end of the office visit if they choose to participate. Baseline demographic information and past medical history including current medications and medications previously tried will be collected. Patients and assessors will not be blinded to treatment.

When the patient is admitted to the hospital for treatment, the neurology team will be the admitting team and will consult the Acute Pain Service (APS) for assistance with management of ketamine, which is standard practice when ketamine is used for headache treatment at TJUH. Patients will be admitted for a total of 5 full days from the time of admission until discharge. Adjustments to ketamine infusion will be made according to standard APS protocol and data will be collected by the research coordinator or other study team personnel. A standard 11-point numeric rating scale (NRS) will be used to obtain pain ratings and they will be collected twice daily. A 4-point pain assessment scale (0=none, 1=mild, 2=moderate, 3=severe) will also be used. Blood samples will be collected at baseline and at 24 hours, 72 hours, and the final day of treatment. They will be performed at external laboratories. A daily headache diary will be used for all patients and they will be given instructions how to use one prior to discharge. A depression screening will be performed on day of admission to TJUH.

Follow-up office visits at approximately 2 weeks and 2 months will be used for collection of pain ratings and medication use. Headache diaries will be collected. If telephone visits occur, assessments will be done over the phone in place of an office visit.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age 18 years and older) who meet the criteria of refractory chronic migraine as defined by the International Classification of Headache Disorders-II definition who present to the Jefferson Headache Center after failing an inpatient course of treatment at Methodist.

Exclusion Criteria:

* Schizophrenia
* active psychosis
* pregnancy
* poorly controlled cardiovascular disease
* cirrhosis
* previous treatment with intravenous ketamine

These criteria are all consistent with the 2018 Consensus Guidelines for Ketamine. Patients who are deemed poor candidates for ketamine by a study team member for any reason, such as intolerance of prior neuroleptic medications, may be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
The improvement in pain after ketamine (0 to 10 numerical rating scale) will be compared to improvement after initial inpatient treatment. | 1 year
  Each patient will serve as his or her own control.
Improvement in a 0-3 qualitative scale where 0=none, 1=mild, 2=moderate, 3=severe pain will be used comparing change from beginning to end of ketamine treatment to change after initial inpatient treatment. | 1 year
  Each patient will serve as his or her own control.

SECONDARY OUTCOMES:
Incidence of adverse effects | 1 year
  The number and severity of adverse effects, including hallucinations, nightmares, nausea/vomiting, blurry vision, sedation, and changes in liver function tests, will be recorded.
Ketamine metabolite levels | 1 year
  Levels of ketamine metabolites, including norketamine, hydroxynorketamines, hydroxyketamines, and dehydronorketamines, will be measured at baseline, 24 h, 48 h, 72 h, and just before infusion is stopped.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Schwenk ES, Dayan AC, Rangavajjula A, Torjman MC, Hernandez MG, Lauritsen CG, Silberstein SD, Young W, Viscusi ER. Ketamine for Refractory Headache: A Retrospective Analysis. Reg Anesth Pain Med. 2018 Nov;43(8):875-879. doi: 10.1097/AAP.0000000000000827. PMID 29923953
- [Background] Cohen SP, Bhatia A, Buvanendran A, Schwenk ES, Wasan AD, Hurley RW, Viscusi ER, Narouze S, Davis FN, Ritchie EC, Lubenow TR, Hooten WM. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Chronic Pain From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):521-546. doi: 10.1097/AAP.0000000000000808. PMID 29870458
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Schulman E. Refractory migraine - a review. Headache. 2013 Apr;53(4):599-613. doi: 10.1111/head.12047. Epub 2013 Feb 13. PMID 23405959
- [Background] Afridi SK, Giffin NJ, Kaube H, Goadsby PJ. A randomized controlled trial of intranasal ketamine in migraine with prolonged aura. Neurology. 2013 Feb 12;80(7):642-7. doi: 10.1212/WNL.0b013e3182824e66. Epub 2013 Jan 30. PMID 23365053
- [Background] Pomeroy JL, Marmura MJ, Nahas SJ, Viscusi ER. Ketamine Infusions for Treatment Refractory Headache. Headache. 2017 Feb;57(2):276-282. doi: 10.1111/head.13013. Epub 2016 Dec 27. PMID 28025837